CLINICAL TRIAL: NCT04461444
Title: COhort for Bardet-Bield Syndrome and Alström Syndrome for Translational Research Etude Interventionnelle Monocentrique
Brief Title: COhort for Bardet-Bield Syndrome and Alström Syndrome for Translational Research Monocentric Interventional Study
Acronym: COBBALT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 7076
Record Dates: First submitted 2019-01-21; First posted 2020-07-08 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Bardet-Biedl Syndrome; Alström Syndrome
MeSH Terms: conditions — Bardet-Biedl Syndrome; Alstrom Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group ALMS et BBS (Other)
  Interventions: Genetic: Skin biopsy

INTERVENTIONS:
Genetic: Skin biopsy — COBBALT is considered as an interventional with minor associated risks and constrains study due to the presence of skin biopsies that may not all be part of the usual medical practice. Risks are those linked to the biopsy procedure:
  * risk of pain due to the procedure performed under local anaesthesia
  * can leave a visible scar (about 2 x 1 cm)

SUMMARY:
ALMS and BBS syndromes are rare diseases with overlapping features of multiple sensory and metabolic impairments, including diabetes mellitus. There are to date no specific treatments available and limited information on the natural history of the diseases. the investigators aim to establish a French cohort for these diseases to improve patient care and assess the effect of actual therapies on quality of life.

The purpose of this study is to establish a cohort of Bardet-Bield syndrome (BBS) and ALström syndrome (ALMS) patients in order to formalize and address questions concerning the in-depth natural clinical and biological history of the disease on the long term for a given patient, establish the impact on the quality of life of various clinical manifestations

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sex
* Age minimum*
* patients with social protection
* Written informed consent form signed prior initiating any trial related procedure:

  * by > 18-year old patients
  * by both parents for minor patients > 4 months or legal representative for protected adults, and by minor and protected adults patients if able to understand and/or give their assent.
  * For foreign patients, a third party will translate, if required, the information prior to the consent.
* a diagnosis of BBS or ALMS based on molecular assessment or clinical evaluation/or patient with mutation and none of the diagnosis criteria
* and/or an identified mutation in BBS genes or ALMS1 gene

  * The inclusion of children is essential to a cohort study that is attempting an early identification of visual, metabolic and renal abnormalities. Many of the age-dependent manifestations of BBS develop during childhood and the average age of diagnosis is 9.2 years

Exclusion Criteria:

* Serious active intercurrent pathology that may impact the collected data
* Patient under judicial protection
* Participation in another interventional clinical trial which includes an exclusion period
* Non protected adult with difficulty of comprehension, or inability to understand the delivered information (emergency situation ...).

Min Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2020-06-16 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2035-02 (Estimated)

PRIMARY OUTCOMES:
Clinical history description of Bardet-Biedl (BBS) and ALström syndromes (ALMS). | 5 years
  renal function, eyes, endocrine, Clinical Examination
Clinical history description of Bardet-Biedl (BBS) and ALström syndromes (ALMS). | 5 years
  Record of biological results
Clinical history description of Bardet-Biedl (BBS) and ALström syndromes (ALMS). | 5 years
  Record of Social Life with questionnaire
Clinical history description of Bardet-Biedl (BBS) and ALström syndromes (ALMS). | 5 years
  Record of treatments (therapy and surgery)

CONTACTS AND LOCATIONS:
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided